CLINICAL TRIAL: NCT02983162
Title: Is the Weighted Genetic Risk Score Associated With Dupuytren Disease Recurrence?
Brief Title: Is wGRS Associated With DD Recurrence?
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, D.C. Broekstra, MSc, University Medical Center Groningen
Other Study IDs: 201600670
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Dupuytren Contracture
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Retrospectively reviewing the participants of the GODDAF database, revealed a significant association between the weighted genetic risk score and Dupuytren disease recurrence. However, a significant dose-response relation was not found. This might be caused by underestimating the recurrence rate, due to the retrospective nature of determining recurrence. Therefore, we want to do a follow-up measurement of the GODDAF participants, to see whether they suffered from recurrent disease.

Objective: We aim to determine whether the wGRS is associated with recurrent DD.

Study design: An observational study, in which the participants of the GODDAF study are followed up.

Study population: Patients affected by Dupuytren disease, aged 18-96 years, who were previously included in another study on the genetic basis of Dupuytren disease.

Intervention (if applicable): NA Main study parameters/endpoints: The main study parameter is the presence of recurrent Dupuytren disease.

ELIGIBILITY:
Inclusion Criteria:

* DD patient
* participant in the GODDAF study
* genetic data passed the quality control
* surgical treatment of DD
* written informed consent

Exclusion Criteria:

* Decisionally incapacitated
* Patients treated for DD with collagenase or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are selected among those who participated in a previous study on the genetic basis of Dupuytren disease (GODDAF). In this study, patients with Dupuytren disease, Peyronie disease or Ledderhose disease and their family members were included. To answer the current research question, only the DD patients are required. The GODDAF study was a multi-center study. For practical reasons, we only want to include patients who were admitted to the UMCG.
  1098 participants were included in the GODDAF study in the Netherlands. Of them 797 were DD patients. Of these 797 patients, we estimate that approximately 85% (677) were admitted to the UMCG. These patients will be approached for participation.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Presence of recurrent Dupuytren disease | 1 day
  there is only one measurement in this study

SECONDARY OUTCOMES:
Severity of Dupuytren recurrence | 1 day
  there is only one measurement in this study

CONTACTS AND LOCATIONS:
Overall Officials: P. MN Werker, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, dept Plastic Surgery, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No